CLINICAL TRIAL: NCT06238206
Title: What User-requirements Need to be Considered When Developing a Lower-limb Exoskeleton? A Qualitative Study.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vrije Universiteit Brussel (Other)
Responsible Party: Principal Investigator, Eva Swinnen, Prof. dr., Vrije Universiteit Brussel
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: RevalEXO1
Record Dates: First submitted 2023-12-13; First posted 2024-02-02 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Stroke; Sarcopenia
Keywords: Assistive technology; Exoskeleton; User perspective; Stroke; Sarcopenia
MeSH Terms: conditions — Stroke; Sarcopenia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- People post-stroke (Experimental): The focus group discussion will assess the needs and requirements of this group.
  Interventions: Other: Focus group discussion
- Older adults with sarcopenia (Experimental): The focus group discussion will assess the needs and requirements of this group.
  Interventions: Other: Focus group discussion
- Physiotherapists (Experimental): The focus group discussion will assess the needs and requirements of this group.
  Interventions: Other: Focus group discussion

INTERVENTIONS:
Other: Focus group discussion — The participant will be asked to take part in three separate focus group discussions implementing the co-design principle. Following the co-design principle the participants will actively contribute towards the primary outcomes. Open questions will be asked to guide the discussion. Interaction between participants will be encouraged.

SUMMARY:
The goal of this study is to identify the needs and requirements of end-users regarding the implementation of a lower-limb exoskeleton in a remote home setting. The end-users include older adults with sarcopenia, post-stroke individuals and physiotherapists. The main question it aims to answer is:

• What are the needs and requirements of the end-user population when developing a lower-limb exoskeleton that can be implemented in a remote home setting?

Participants will engage in three separate focus group sessions, in which they will discuss the predetermined topics. Interactions between the participants will be guided by open questions.

ELIGIBILITY:
People post-stroke:

Inclusion Criteria:

* > 18 years old
* ≥ 3 months ago stroke diagnosis
* Current difficulties during gait

Exclusion Criteria:

* Serious speech disorder
* Lowered cognitive competence

Older adults with sarcopenia:

Inclusion Criteria:

* > 65 years old
* Difficulties during chair sit to stand
* Current difficulties during gait

Exclusion Criteria:

* Lowered cognitive competence

Physiotherapist:

Inclusion Criteria:

* Currently active as a physiotherapist
* Experience in treating people with sarcopenia and/or post-stroke conditions

Exclusion criteria:

* Can't verbally answer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2024-01-17 (Actual); Primary Completion 2024-04-05 (Actual); Study Completion 2024-04-05 (Actual)

PRIMARY OUTCOMES:
User Personas | 8 weeks
  A set of personas (=representation of a group of individuals with common characteristics) will be defined for both the older adults with sarcopenia and the stroke survivors. This is identified through the qualitative analysis of the answers on predefined open questions during the focus group discussion.
Identification of Activities for Exoskeleton Use | 8 weeks
  Specific activities where exoskeletons demonstrate added value will be defined. This is identified through the qualitive analysis of the answers on predefined open questions during the focus group discussion.
Interface and Design Concept Formulation | 8 weeks
  Key elements on the interface and design concept of exoskeletons will be described. This is identified through the qualitive analysis of the answers on predefined open questions during the focus group discussion.
Digital Rehabilitation Outcomes | 8 weeks
  Key elements of rehabilitation measures that an exoskeletons should be able to assess will be described. This is identified through the qualitive analysis of the answers on predefined open questions during the focus group discussion.

CONTACTS AND LOCATIONS:
Overall Officials: Eva Swinnen, PhD, Principal Investigator — Vrije Universiteit Brussel
Locations (1):
- Brubotics Rehabilitation Research Center, Jette, Brussels Capital, Belgium